CLINICAL TRIAL: NCT04673253
Title: Can Passive Leg Raise Prevent Spinal Anesthesia-induced Hypotension During Cesarean Section?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Ozyurt, Medical Doctor, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AntalyaEAH03
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Hypotension
Keywords: cesarean section; hypotension; spinal anesthesia; passive leg raise
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive leg raise (Active Comparator): group for passive leg raise
  Interventions: Other: Passive leg Raise
- Control (Placebo Comparator)
  Interventions: Other: control

INTERVENTIONS:
Other: Passive leg Raise — The intervention will be performed immediately after spinal anesthesia, and passive leg raise will be performed using two standard pillows placed under the heel so that the leg is approximately 30 cm above the horizontal plane of the table. The passive leg raising position will continue until the cord is clamped.
  Arms: Passive leg raise
Other: control — The controlled group was positioned in the normal supine position.
  Arms: Control

SUMMARY:
All over the world, spinal anesthesia is widely used in cesarean sections due to its superiority over general anesthesia. Due to reasons such as increased sensitivity to local anesthetics and increased intra-abdominal pressure in pregnant women, the frequency of hypotension increases by up to 70%. As a result of the blockage of sympathetic vasoconstrictor fibers originating from T1-L2 segments, loss of peripheral resistance, venous ponding occurs, and cardiac output decreases. Also, the level required for cesarean operation is T4 or T5, and the possibility of affecting the cardiac accelerator fibers, so bradycardia due to the increase in parasympathetic activity may deepen the hypotension. If postspinal hypotension is not managed correctly, it may lead to maternal and fetal complications. In addition to classical methods such as fluid loading and prophylactic vasoconstrictor application to prevent hypotension in pregnant women after spinal anesthesia, techniques such as wrapping the lower extremity, lifting, or applying both together have been in question.

Passive leg raise application is an easy method that allows the blood collected in the lower part of the body to participate in the central circulation with the effect of gravity. An increase in venous return occurs with the passage of blood from the lower extremities to the thorax. Thus, it leads to an increase in stroke volume and an increase in cardiac output. In this study, we aimed to determine the effectiveness of passive leg raising in preventing or reducing the depth of hypotension after spinal anesthesia in pregnant women who underwent cesarean section under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Parturients who are planned for the elective cesarean section

Exclusion Criteria:

* Failed spinal block
* Shift to general anesthesia
* Severe cardiac disease
* Hypertensive disorders of pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Before the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 1 minute after the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 2 minutes after the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 3 minutes after the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 4 minutes after the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 5 minutes after the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 7 minutes after the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 9 minutes after the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 11 minutes after the spinal anesthesia in the supine position
  Systolic blood pressure will be recorded from the monitor
Systolic blood pressure | 1 minute after the umblical cord clamping
  Systolic blood pressure will be recorded from the monitor

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No